CLINICAL TRIAL: NCT03461328
Title: Effect of Intravenous Infusion of Magnesium Sulphate on Arterial Oxygenation and Pulmonary Mechanics in Patients With Chronic Obstructive Pulmonary Diseases Undergoing Cancer Larynx Surgery. A Randomized Controlled Trial
Brief Title: Effect of Magnesium Sulphate Infusion on Lung Mechanics and Oxygenation in COPD Patients Undergoing Total Laryngeal
Acronym: COPD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Abeer Ahmed, MD, Assistant Professor of Anesthesia and SICU - Faculty of Medicine - Cairo University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: N-76-2017
Record Dates: First submitted 2018-02-20; First posted 2018-03-12 (Actual); Last update posted 2019-08-21 (Actual); Status verified 2019-08

CONDITIONS: Chronic Obstructive Pulmonary Diseases
Keywords: magnesium sulphate, chronic obstructive pulmonary diseases
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Magnesium Sulfate

STUDY DESIGN:
Intervention Model Description: Intra-operative intravenous infusion of magnesium sulphate in patients with chronic obstructive pulmonary diseases undergoing total laryngectomy and assess the influence on arterial oxygenation and pulmonary Mechanics in
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mg-group (Experimental): 10% MgSO4 solution will be used, a loading dose of 30mg/kg over 20 min (equivalent to infusion rate of 0.9 ml/kg/hr for 20 min) will be given followed by continuous infusion of 10mg/kg/hr (equivalent to infusion rate of 0.1ml/kg/hr).
  Interventions: Drug: Magnesium Sulphate
- Control group (No Intervention): In control group, same rates of infusion for loading and maintenance will be applied using 0.9 normal saline.

INTERVENTIONS:
Drug: Magnesium Sulphate — intra-operative infusion of of 10% MgSO2 , stating by a laoding dose of 30be used, a loading dose of 30 mg/kg over 20 min followed by continuous infusion of 10 mg/kg/hr accomplish the total laryngectomy.
  Arms: Mg-group

SUMMARY:
Chronic Obstructive Pulmonary Disease [COPD] is a major cause of chronic morbidity and mortality worldwide. COPD is characterized by persistent progressive airflow limitation that adversely affects the ventilation/perfusion (V/Q) matching and mechanics of the respiratory muscles and leads to hypoventilation and reduced gas transfer. COPD was identified as a significant comorbidity associated with increased incidences of postoperative pulmonary complications and prolonged hospital stay. MgSO4 either intravenous or inhalational has been shown to promote bronchodilation and to improve lung function in asthmatic patients. MgSO4 either intravenous or inhalational has been shown to promote bronchodilation and to improve lung function in asthmatic patients. Administration of MgSO4 in patients with stable COPD was associated with reduced lung hyperinflation and improvement of respiratory muscle strength. This randomized control trial is designed to assess the effect of intravenous MgSO4 infusion on oxygenation and pulmonary mechanics and incidence of postoperative pulmonary complications and length of hospital stay in patients with COPD undergoing cancer larynx surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing cancer larynx surgery (partial laryngectomy, total laryngectomy with or without neck dissection).
* Age more than 40 years old
* ASA physical status II and III.
* Diagnosed as having COPD by preoperative spirometry. The classification is bases on the post-bronchodilators forced expiratory volume in the first second (FEV1). Mild COPD is diagnosed when FEV1 is > 80% of predicted while moderate COPD is diagnosed when FEV1 is < 80% and > 50% of predicted and sever COPD is diagnosed when FEV1 is < 50% and > 30% of predicted

Exclusion Criteria:

* o Patients with heart failure.

  * History with arrhythmias or treatment with antiarrhythmic drugs.
  * Patient with heart block or on beta blockers or calcium channel blockers.
  * Patients with impaired renal function (creatinine > 2)
  * Patients with impaired liver function (ALT more than 2 folds).
  * Patient with combined restrictive and obstructive pulmonary disease.
  * Patients with preoperative tracheostomy.
  * Patients with huge mass obstructing > 50% of the view. (due to its influence on the spirometry measurements).

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-04-20 (Actual); Primary Completion 2018-10-20 (Actual); Study Completion 2019-03-20 (Actual)

PRIMARY OUTCOMES:
lung oxygenation | over a period of 6-8 hours, from the time of induction of general anesthesia until time of patients discharge from the PACU.
  PaO2/FiO2 immediately after arrival to the PACU

CONTACTS AND LOCATIONS:
Locations (1):
- Anesthesia department - Faculty of medicine- Cairo University, Cairo, Egypt

REFERENCES:
- [Derived] Ahmed A, Sayed AH, Elkholy J, Elshal S, Badwy A, Abdelhamid B, Ollaek M. Intraoperative MgSO4 infusion protects oxygenation and lung mechanics in COPD patients during general anesthesia. A randomized clinical trial. Acta Anaesthesiol Scand. 2020 Nov;64(10):1460-1468. doi: 10.1111/aas.13684. Epub 2020 Aug 16. PMID 32770840